CLINICAL TRIAL: NCT00828438
Title: A Phase 1, Open-Label, Single-Dose Study of the Pharmacokinetic Properties of Lorcaserin in Subjects With Renal Impairment
Brief Title: Pharmacokinetic Properties of Lorcaserin in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APD356-016
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2009-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lorcaserin 10mg (Experimental)
  Interventions: Drug: Lorcaserin 10mg

INTERVENTIONS:
Drug: Lorcaserin 10mg

SUMMARY:
The purpose of this study is to evaluate the PK properties of lorcaserin in subjects with end stage renal disease (ESRD) who require dialysis and will be studied under dialysis and non-dialysis conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged between 18 and 79 years (inclusive)
2. Able to give signed informed consent
3. Renal function will fall into one of the following categories (ideal body weight will be used for the calculation):

   * One-fifth of subjects will have normal renal function, defined as creatinine clearance > 80 mL/min calculated using the Cockroft-Gault equation
   * One-fifth of subjects will have creatinine clearance 51-80 mL/min
   * One-fifth of subjects will have creatinine clearance 31-50 mL/min
   * One-fifth of subjects will have creatinine clearance 5-30 mL/min, but not require dialysis
   * One-fifth of subjects will have chronic end stage renal disease, require regularly scheduled hemodialysis, and be on a stable hemodialysis regimen for at least 3 months prior to dosing
4. Subjects in the renally impaired groups will have stable renal disease as per Investigator's assessment, with no clinically meaningful changes for 1 month prior to randomization.
5. Subjects in all groups will have a BMI of 27-45 kg/m2.
6. Considered to be in stable health in the opinion of the Investigator.
7. Eligible male and female subjects must agree not to participate in a conception process.

Exclusion Criteria:

1. Prior participation in any study of lorcaserin.
2. Clinically significant new illness in the 1 month before screening
3. Not suitable to participate in the study in the opinion of the Investigator including an existing physical or mental condition that prevents compliance with the protocol
4. History of any of the following cardiovascular conditions:

   * Myocardial infarction (diagnosed by cardiac enzyme[s] and/or diagnostic ECG), CVA, TIA or RIND within 3 months of screening
   * Cardiac arrhythmia requiring initiation of a new medical or surgical treatment within 3 months of screening (pacemaker and/or defibrillator implanted > 3 months prior to screening is acceptable)
   * Unstable angina
   * History of pulmonary artery hypertension
5. Positive result of HIV, hepatitis B or hepatitis C screens.
6. Malignancy within 2 years of the screening visit (except basal cell or squamous cell carcinoma with clean surgical margins)
7. Use of SSRI's, SNRI's, and other medications must meet washout period.
8. Recent history (within 3 months prior to the screening visit) of alcohol or drug/solvent abuse or a positive screen for drugs of abuse at screening.
9. Participated in any clinical study with an investigational drug, biologic, or device within 1 month prior to dosing
10. Unwilling, or whose partner is unwilling, to use an adequate means of contraception during and for 1 month following completion/withdrawal of the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the pharmacokinetic properties of lorcaserin in subjects with mild, moderate or severe renal impairment as compared to subjects with normal renal function.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of lorcaserin in subjects with renal impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

REFERENCES:
- [Derived] Christopher RJ, Morgan ME, Tang Y, Anderson C, Sanchez M, Shanahan W. Pharmacokinetics and Tolerability of Lorcaserin in Special Populations: Elderly Patients and Patients with Renal or Hepatic Impairment. Clin Ther. 2017 Apr;39(4):837-848.e7. doi: 10.1016/j.clinthera.2017.03.004. Epub 2017 Mar 30. PMID 28365033